CLINICAL TRIAL: NCT02769949
Title: Evaluation of Patients With Genetic Disorders
Brief Title: Pediatric Patients With Metabolic or Other Genetic Disorders
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160103; 16-CH-0103
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-09-24

CONDITIONS: Genetic Disorder; Asperger Disorder; Autism Spectrum Disorder; Fragile X Syndrome; Developmental Delay
Keywords: Genetics; Metabolic; Dysmorphic Syndromes; Developmental Delay; Genetic Counseling; Natural History
MeSH Terms: conditions — Genetic Diseases, Inborn; Asperger Syndrome; Autism Spectrum Disorder; Fragile X Syndrome; Learning Disabilities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family members: Family members (adult and pediatric; affected and unaffected) may be enrolled for the purpose of determining the molecular lesion(s) responsible for genetic disorders.
- Genetic disorders: Participants with genetic disorders

SUMMARY:
Background: Some patients with unusual genetic conditions are referred to the National Institutes of Health (NIH). They may not be eligible to join current research studies. Testing such patients is a good way to improve the skills of research staff. The findings could lead to new processes and research.

Objectives:

To recruit a diverse group of pediatric subjects with genetic disorders. To give clinic staff hands-on experience working with these patients.

Eligibility:

Children any age with a known or suspected genetic disorder.

Design:

Participants will be screened with medical history and physical exam. They may have lab and other tests.

Family members may give DNA samples.

Participants will have:

Medical history

Physical exam

Height, weight, and other measurements taken.

A clinical evaluation of their disorder.

They may have:

Blood, urine, and saliva samples taken

Imaging tests. These may include x-rays, scans, ultrasound, or skeletal survey.

A sleep study

A visit with other specialists at NIH

A genetic test from a commercial lab

Medical photographs taken

Other tests

Participants may have follow-up visits. They may get medical or surgical treatment.

DETAILED DESCRIPTION:
The aim of this protocol is to allow genetic-related evaluations for patients with a variety of known or suspected genetic disorders.) If not eligible for a specific NICHD research protocol, patients with genetic-related conditions may be evaluated under the auspices of this protocol to provide stimuli for new clinical research initiatives. Standard medically-indicated laboratory or radiological studies may be performed to confirm a diagnosis or to aid in the management of the patient. Clinical data and excess biospecimens collected as part of clinical care will be analyzed for research purposes. In some cases, the subjects may receive medical or surgical treatment for their disorder at the NIH CC according to current clinical practice. The overall purpose of genetic evaluations under this protocol is to support our research missions, generate hypotheses bank specimens for analysis or future use as controls. Family members of subjects evaluated on this protocol (who have informative meiotic inheritance relationships to the proband or index case) may also be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects of any age with known or suspected genetic disorder
* For relatives of subjects with a genetic disorder: Subject is a family member of the proband

EXCLUSION CRITERIA:

-Presence of a medical, psychiatric, or social condition which, in the opinion of the investigator, would place undue burden on the subject, NIH resources, or increase risk of participation

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community dwelling participants with genetic disorders
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Recruit Patients with Suspected or diagnosed genetic diseases | Ongoing
  observational/exploratory suspected or diagnosed genetic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Abdennadher M, Inati SK, Rahhal S, Khan O, Bartolini L, Thurm A, Theodore W, Miller JS, Porter FD, Bianconi S. Characterization of seizures and EEG findings in creatine transporter deficiency due to SLC6A8 mutation. Am J Med Genet A. 2024 Feb;194(2):337-345. doi: 10.1002/ajmg.a.63418. Epub 2023 Oct 18. PMID 37850681
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CH-0103.html